CLINICAL TRIAL: NCT03306745
Title: Micronutrient Supplementation for Women With PCO-syndrome - Influence of Nutrition and Physiology on the Development of PCOS-typical Parameters
Brief Title: Micronutrient Supplementation in PCO-syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Johannes Ott, Assoc.-Prof. Priv.-Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1232/2016
Record Dates: First submitted 2017-07-16; First posted 2017-10-11 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Polycystic Ovary Syndrome; Infertility, Female; Micronutrient Deficiency
Keywords: Polycystic Ovary Syndrome; Anti-Mullerian Hormone; Androgens; Micronutrient Supplementation
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility, Female | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The medications are unlabeled for both groups and will be dispensed in unlabeled blisteres. However, patients could search for the actual look of the PROfertil ® female soft capsules and the pills (for example on the internet). Since they differ from the folic acid capsules, patients could identify the control medications. We are aware of the fact that this kind of blinding is not according to standards and could introduce some kind of bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): * 1 soft capsule/day containing 500mg omega-3 fatty acids
  * one tablet/day containing 800mg folic acid, 70mg selenium, 30 mg Vitamin E, 4 mg catechin, 12 mg glycyrrhizin, and 30 mg coenzyme Q10
  Interventions: Dietary Supplement: Profertil female
- Control group (Placebo Comparator): 200µg folic acid - two capsules per day
  Interventions: Dietary Supplement: Folic acid 400 mg

INTERVENTIONS:
Dietary Supplement: Profertil female — For micronutrient ingredients please see details above. PROfertil ® female is approved in Austria by the Austrian Ministry of Health and has a "Free Sales Certificate".
  Arms: Study group
Dietary Supplement: Folic acid 400 mg — Folic acid 400 mg
  Arms: Control group

SUMMARY:
The role of micronutrients in fertility has recently gained increased attention. In women who suffer from polycystic ovary syndrome (PCOS) and infertility, we aim to test the impact of a standardized, multinutrient supplementation on the course of PCOS-specific parameters namely anti-Mullerian hormone (AMH), testosterone, and androstenedione. A total of 60 infertile women with PCOS, previously untreated, will be randomized to receive either a combined standardized multinutrient supplementation (containing folic acid, selenium, vitamin E, catechins, glycyrrhizin, coenzyme Q10 and omega-3-fatty acids; study group) or folic acid alone (control group) in a double-blinded, randomized manner. These study medications will be provided for 3 months and pre- to posttreatment levels of AMH, testosterone, and AMH will be analysed. The study will be performed at the Clinical Division of Gynecologic Endocrinology and Reproductive Medicine of the Medical University of Vienna.

DETAILED DESCRIPTION:
Introduction and scientific background:

In the Western world, malnutrition and subfertility have become increasingly common problems affecting both men and women. A recent study showed that conforming to nutritional recommendations significantly increased the probability of a clinical pregnancy following vitro fertilisation (IVF)/ intracytoplasmatic sperm injection (ICSI). They included fruit, vegetables, certain types of meat, fish, whole-grain products and specific fats (according to the Netherlands Nutrition Centre Foundation). Another study specifically analysed preconceptional consumption of unsaturated fatty acids by women before IVF/ICSI. It discovered a positive effect on the embryo's morphology.

The effect of micronutrients on female fertility is currently under investigation. A 2012 review on the subject included 13 studies with more than 90,000 female participants and provided no generalised recommendations, but allowed the authors to deduce a certain positive effect of supplementation with certain micronutrients on female fertility.

This current study will test the effect of a currently available micronutrient supplementation in women suffering from polycystic ovary (PCO)-syndrome and sterility. The product (PROfertil ® female, Lenus Pharma, Seeböckgasse 59, 1160 Vienna, Austria) is based on several studies that showed (i) an increased need for these micronutrients of women with a desire to have a child or currently pregnant and/or (ii) a positive effect on female fertility. PROfertil ® female is a micronutrient supplement containing selenium, vitamin E, catechins, glycyrrhizin, co-enzyme Q10, folic acid and omega-3 fatty acids.

This study seems of impact from a scientific perspective. Clinical experience with PROfertil ® female suggests that patients suffering from PCO-syndrome experience an increase of anti-müllerian hormone and androgen levels. The reductive effect of PCO-typical serum parameters can be explained pathophysiologically: A chronic low-level pro-inflammatory state - both locally in the ovary and systemically - appears to be among the central pathophysiological correlates of PCO-syndrome. PROfertil ® female contains a mix of several antioxidative agents. A favourable effect on PCO-syndrome is expected. Metformin is an anti-inflammatory substance commonly used to treat PCO-syndrome. The anti-inflammatory effect is seen as positive. This explains why women suffering from PCO-syndrome without insulin-glucose balance problems react positively to treatment with metformin.

The aim of this study is to perform a prospective randomized test comparing PROfertil ® female to supplementation with folic acid alone for female patients suffering from PCO-syndrome and infertility. Supplementation with folic acid is the current state of the art in micronutrient supplementation of infertile women.

Study aims The primary aim of this study is to analyse the effects of three months of treatment with PROfertil ® female compared to a supplementation with 400µg of folic acid for women suffering from PCO-syndrome, sterility, anovulation. The study will examine the parameters typical for PCO-syndrome (anti-müllerian hormone, total testosterone, androstenedione).

The secondary goal is to document the individual course of further fertility treatment.

The products being administered to the patients for four weeks are:

* PROfertil ® female (Lenus Pharma Gesellschaft mit beschränkter Haftung [GesmbH], Seeböckgasse 59, 1160 Vienna; treatment group) - one soft capsule (500mg Omega-3-fatty acids) and one pill (folic acid: 800µg, selenium 70µg, vitamin E 30mg, catechine: 4mg, glycyrrhizin 12mg, and coenzyme Q10: 30mg) per day.
* 200µg folic acid (folic acid capsules 400µg ®, OTC Produktion und Forschung GesmbH, Fischergasse 17, 5020 Salzburg; control group) - two capsules per day.

The study will be performed in a double-blinded manner. The medications are unlabeled for both groups and will be dispensed in unlabeled blisters. However, patients could search for the actual look of the PROfertil ® female soft capsules and the pills (for example on the internet). Since they differ from the folic acid capsules, patients could identify the control medications. The study team is aware of the fact that this kind of blinding is not according to standards and could introduce some kind of bias.

Study hypotheses:

First hypothesis: A three-month treatment with PROfertil ® female causes a drop of anti-müllerian hormone, total testosterone and androstenedione levels. This does not happen if treated with 400µg folic acid.

Outcome parameters:

Primary outcome parameters: anti-müllerian hormone (AMH), total testosterone and androstenedione levels

Study design:

Monocentric, prospective randomized double-blinded trial

Recruitment:

The participants are recruited by medical professionals at the Department of Obstetrics and Gynecology of the Medical University of Vienna using the above mentioned criteria during routine examinations before any treatment for PCO-syndrome and/or sterility is initiated. Potential participants are informed about the procedure, clinical relevance and possible additional effort caused by study participation. The patients willing to participate then have to sign the written informed consent.

Sample size calculation:

Assuming a reduction of the mean AMH levels by 2 ng/ml at a standard deviation of 3 ng/ml and an alpha value of 0.05 and a power of 0.90, the paired t-test requires 26 patients per group. Due to the fact that the participants wish to conceive a child and have been diagnosed with sterility, a low drop-out rate can be expected. There is no reliable data on this or similar treatments that allow prediction of the chance to conceive. Due to the favourable benefit-to-risk profile, a 15% drop-out rate is assumed. This corresponds to 4 patients per group. Thus, the final sample size is calculated as 30 patients per group, which leads to a total study population of 60.

Statistical analysis:

The bio-statistician will randomise the data using nQuery advisorTM Version 7.0. The information will then be packaged in an envelope by a person independent of the participating medical professionals and other scientific personnel. This will only be opened after the inclusion of the patient. Categorical variables will be presented as absolute numbers and percentages, numerical variables as median and interquartile range.

The following statistical analyses are planned: The result parameters and the patient characteristics of the two groups will be compared using the Welch test (for numerical variables) and the Chi-square-test or Fisher's exact test (for categorical variables). A p-value of <0.05 is considered to be statistically significant. The statistical analyses will be performed using SPSS 24.0 for Windows (SPSS Inc, 1989-2017).

Further details on study design:

After recruiting the participants at the outpatient clinics for Gynecologic Endocrinology and Infertility Treatment, they are randomly assigned to one of the groups.

Participants will receive either 2 unlabelled soft capsules containing 200µg folic acid each or 1 unlabelled soft capsule containing omega-3 fatty acids and 1 tablet containing folic acid, selenium, vitamin E, catechins, glycyrrhizin, and co-enzyme Q10 (see Table above for details on doses).

The planned examination of AMH, total testosterone and androstenedione levels will take place after a minimum of 90 days (and a maximum of 100 days) after beginning supplementation with PROfertil ® female or folic acid. The maximum duration of participation is thus 100 days. After taking the micronutrient supplementation (PROfertil ® female or folic acid) beyond the planned minimum treatment duration, an individualised fertility treatment can be performed.

There are two study-specific consultations: After including the patient (consultation 1: randomisation, distribution of drugs and start of study) and after 90 to 100 days (consultation 2). During consultation 2, unused study blisters are collected and patients are questioned on peculiarities and possible side effects of the micronutrient supplementation used.

It is expected that 30 minutes for consultation 1 and 15 minutes for consultation 2 will have to be spent by the patient. The consultations will be held during regular outpatient treatments and will be part of the planned routine examinations. They include discussions of examination results and recommendations for further treatment.

Benefits-to-risk assessment and preventive measures:

Risks or complications due to the use of PROfertil ® female and additional venepuncture are not expected. A recent study using the same product showed no substance-related side effects (number of the ethics committee of the Medical University of: 1659/2013; accepted on 2013-09-24) (9). A direct benefit for the treatment group is possible. A positive effect on PCO syndrome can be assumed, which might result in a higher chance of pregnancy. The substance administered to the control group is state of the art for female fertility treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has been diagnosed with PCO-syndrome using revised 2004 Rotterdam-criteria (7).
2. The patient is sterile, defined as being unable to become pregnant within a year despite unprotected sexual intercourse.
3. The patient suffers either from oligomenorrhoea (defined as an interval of ≥60 days between the last three menstruations) or complete amenorrhoea for at least 90 days.
4. The patient has given her written informed consent after detailed information on the study by medical professionals at the Department of Obstetrics and Gynecology of the Medical University of Vienna.
5. Both partners are at least 19 years old and are younger than 35. The age limit was chosen to take physiologically reduced fertility beyond this age (8). This measure allowed the women to avoid a 100-day delay of fertility treatments due to this study.

Exclusion Criteria:

1. No informed consent.
2. At least one partner is younger than 19 years or older than 35 years.
3. The patient has been subject to one of the following PCO-syndrome-related treatments within three months before inclusion: metformin, combined oral contraceptives, cortisol therapy, inositol, ovarian drilling, any kind of ovarian stimulation, in-vitro fertilisation. Promoting menstruation using gestagen products is acceptable.

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Anti-Mullerian Hormone (AMH) | Change from pre-treatment, baseline serum level to serum level at 3 months of treatment.
  Change in serum AMH level
testosterone | Change from pre-treatment, baseline serum level to serum level at 3 months of treatment.
  Change in serum testosterone level
androstenedione | Change from pre-treatment, baseline serum level to serum level at 3 months of treatment.
  Change in serum androstenedione level

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Clinical Division of Gynecologic Endocrinology and Reproductive Medicine, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hager M, Nouri K, Imhof M, Egarter C, Ott J. The impact of a standardized micronutrient supplementation on PCOS-typical parameters: a randomized controlled trial. Arch Gynecol Obstet. 2019 Aug;300(2):455-460. doi: 10.1007/s00404-019-05194-w. Epub 2019 May 17. PMID 31101977

DOCUMENTS (2):
  • Study Protocol (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT03306745/Prot_001.pdf
  • Statistical Analysis Plan (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT03306745/SAP_002.pdf